CLINICAL TRIAL: NCT04050852
Title: Pulmonary Function Test Changes and Respiratory Muscle Strength Trends in Spinal Muscular Atrophy Patients Receiving Nusinersen Treatments
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: no enrolled prospects
Sponsor: NYU Langone Health (Other)
Collaborators: Winthrop University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-00242
Record Dates: First submitted 2019-08-07; First posted 2019-08-08 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Spinal Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — nusinersen

STUDY DESIGN:
Intervention Model Description: 5-10 patients with spinal muscular atrophy (SMA), ages 5 years old and above, who have already consented to nusinersen treatment, or have already initiated nusinersen (spinraza) treatments at NYU Winthrop Hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SMA patients receiving nusinersen treatments (Experimental)
  Interventions: Drug: Nusinersen Treatments

INTERVENTIONS:
Drug: Nusinersen Treatments — Antisense oligonucleotide, which targets the SMN2 pre-mRNA, particularly exon 7.
  Other Names: Spinraza

SUMMARY:
It is well known that patients with spinal muscular atrophy (SMA) have progressive decline of respiratory muscle function. Therapy traditionally involved supportive means to ensure optimal nutrition and airway clearance. Nusinersen (spinraza) is a disease-modifying medication approved for treatment of SMA in pediatric and adult patients. The goal of this study is to observe pulmonary function test (PFT) changes and respiratory muscle strength trends throughout the first year of treatment. A prospective, longitudinal study measuring pulmonary function testing (PFTs) changes in spinal muscular atrophy (SMA) patients. Patients will be patients with SMA who are approved and maintained on nusinersen. Patient will have a baseline PFT. Investigators will repeat PFT at 3, 6, and 12 months while on nusinersen treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with SMA of any type who are eligible to start nusinersen treatments at NYU Winthrop Hospital.

Exclusion Criteria:

* Patients unable to comply with nusinersen treatments according to recommended schedule (first 3 doses every 2 weeks, then the 4th dose is administered 1 month after the 3rd dose, and then maintenance dose administered every 4 months).

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
percent improvement Maximum inspiratory pressure (MIP) | 3, 6, and 12 months
  is the pressure developed during forceful inspiration against an occlusion. It is measured at end expiratory phase (near residual volume) and assesses inspiratory muscle strength (diaphragm, external intercostal muscles, and accessory muscles). Normal values for healthy adult females -50 cmH2O and healthy males -75 cmH2O.
percent improvement Maximum expiratory pressure (/MEP) | 3, 6, and 12 months
  the pressure developed during forceful expiration against an occlusion. It is measured at end inspiratory phase (near TLC) and assesses expiratory muscle strength (abdominal muscles, internal intercostal muscles, and accessory muscles). Normal values for healthy adult females +80 cmH2O and healthy males +100 cmH2O.

CONTACTS AND LOCATIONS:
Overall Officials: Melodi Pirzada, MD, Principal Investigator — New York Langone Medical Center
Locations (1):
- NYU Langone Health, New York, New York, United States